CLINICAL TRIAL: NCT04796233
Title: Patient Perspectives on Advance Care Planning Discussions Prior to Cardiac Surgery
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other)
Responsible Party: Sponsor
Other Study IDs: 19-5910
Record Dates: First submitted 2021-03-10; First posted 2021-03-12 (Actual); Last update posted 2021-09-01 (Actual); Status verified 2021-02

CONDITIONS: Cardiac Surgery
Keywords: Advance Care Planning

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The purpose of this study is to explore patient perspectives on Advance Care Planning (ACP) prior to cardiac surgery, including perceptions of benefits, drawbacks, and barriers to ACP.

DETAILED DESCRIPTION:
In this study, we plan to interview 40 patients who are scheduled to undergo cardiac surgery about their perspectives on preoperative ACP and discussion of their values, goals of care, and preferences for prolonged care in hospital prior to having surgery. We plan to conduct and audio record one-on-one interviews that are structured around standard questions about ACP. After recordings are completed, we plan to conduct an analysis of the interviews to find common themes and ideas that participants have about preoperative advance care planning. These results will help us understand whether patients value and wish to participate in advance care planning prior to major surgery, and will help to guide the structure and content of preoperative advance care plan programs in the future.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients undergoing cardiac surgical procedures that involve a sternotomy, thoracotomy, or cardiopulmonary bypass for any indication.
* Age > 18
* English-speaking

Exclusion Criteria:

* Emergency surgery, regardless of indication or procedure
* Minor/percutaneous cardiac procedure
* Lack of decisional capacity due to dementia or other neurocognitive dysfunction
* Previously decided upon advance care directives
* Still considering surgery or not yet booked for an operation

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: We will enroll patients at Toronto General Hospital, a tertiary cardiac surgery centre in Toronto. We will include patients undergoing any cardiac surgery procedures that involve cardiopulmonary bypass, as well as patients undergoing off-pump coronary bypass procedures and any other high-risk cardiac surgery patients, for example, those undergoing ventricular assist device insertion or pericardectomy.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2021-10 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
Interview | 30-35 Minute interview
  Patient perspectives and attitudes regarding advance care planning (ACP) with a focus on patient values and goals prior to cardiac surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Michael Tylee, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Toronto General Hospital - University Health Network, Toronto, Ontario, Canada